CLINICAL TRIAL: NCT04073082
Title: Safety and Efficacy of Er:YAG and Nd:YAG Laser Therapy in Gynecology: A Retrospective Case Series.
Brief Title: Safety and Efficacy of Laser Therapy in Gynaecology
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Juna d.o.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: J01
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Herpes Genitalis; Genital Wart; Lichen Sclerosus; Cervical Intraepithelial Neoplasia; Labial Reduction Surgery; Episiotomy Scar; Bartholin Cyst; Hidradenitis Suppurativa
MeSH Terms: conditions — Herpes Genitalis; Condylomata Acuminata; Lichen Sclerosus et Atrophicus; Uterine Cervical Dysplasia; Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to retrospectively evaluate the effectiveness and safety of Er:YAG laser for treatment of different gynecological indication, e.g. genital lesions, Bartholin's cyst, condyloma, episiotomy scars, lesions of hydradenitis suppurativa and use of laser in genital surgery used in private practice.

ELIGIBILITY:
Inclusion Criteria:

* patients with any of the selected gynecology indications, treated with laser in the period 2013-2018
* signed informed consent

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective study assessing the safety and efficacy of laser use in treatment of different gynecology indications.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-01-24 (Estimated); Study Completion 2020-01-24 (Estimated)

PRIMARY OUTCOMES:
Safety - occurence of adverse effects. | [1 year]
  Recording if any adverse effects occur.
Efficacy - number of laser treatments. | [1 year]
  Number of laser treatments needed for lesion clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Urška Urska.Bizjak-Ogrinc@juna.si, MD, MSc, Principal Investigator — Specialist in obstetrics and gynecology
Locations (1):
- Juna, Ljubljana, Slovenia